CLINICAL TRIAL: NCT01624155
Title: Utilizing the Electronic Medical Record to Collaborate With a Community- Based Organization to Increase More Effective Contraception Utilization Among Women Prescribed Teratogenic Medications
Brief Title: Increasing Contraception Utilization Among Women Prescribed Teratogenic Medications
Acronym: TLC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Christina Chambers, Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 111808
Record Dates: First submitted 2012-06-01; First posted 2012-06-20 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Teratogenesis
Keywords: teratogens; contraception; electronic medical record
MeSH Terms: conditions — Teratogenesis | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The patient is contacted by a specialist in the CTIS Pregnancy Health Information in the Department of Pediatrics at UCSD, and a brief patient interview is conducted with a risk assessment and counseling regarding her medication and the potential effects if she were to become pregnant. The patient is also given information about contraceptive methods, efficacy rates, and the safety of each method based on the USMEC guidance for the patient's medical condition.
  After the counseling is completed, the patient is asked if she is interested in participating in the research study. If the patient consents to participation, she is contacted one week, one month, and three months after the initial telephone interaction and asked several questions regarding her current contraceptive utilization and any changes from the time of the last interview. Upon completion of the three-month follow-up, participants are asked to complete a satisfaction survey.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Women taking teratogens (Experimental): Women taking teratogens
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — EMR referral to teratogen and contraception counseling

SUMMARY:
Typically, the CTIS Pregnancy Health Information Line in the Department of Pediatrics, School of Medicine at the University of California educates pregnant women who call the Information Line after an exposure to a medication that might be harmful to the developing baby has already taken place, and therefore the opportunity for prevention of that exposure no longer exists. Frequently these pregnancies are unintended and occur due to the lack of effective contraceptive use. This study facilitates patient access at UCSD to specialized and individualized contraceptive counseling for women of reproductive age who are currently taking a medication that might be risky in a future pregnancy. This study also measures the impact of individualized contraceptive counseling in changing contraceptive behavior.

Primary Hypothesis: EPIC (EMR)/physician-facilitated referral of female patients of reproductive age to an existing specialized counseling service at UCSD will improve the utilization of more effective contraception among women of reproductive age who are prescribed medications that might be harmful to the developing fetus.

DETAILED DESCRIPTION:
This is a prospective cohort study to evaluate a) the effectiveness of the referral system from Family Medicine to the CTIS Pregnancy Health Information Line, and b) the impact of specialized counseling on contraceptive behavior change among the subset of women who accept the counseling and enroll in the follow-up study.

If a woman of reproductive age is seen by a Family Medicine clinician and she is currently taking or is newly prescribed one of the target medications, an EMR electronic alert will be generated for the clinician. The alert will say "This patient may benefit from a referral to the CTIS Pregnancy Health Information Line for counseling," click "Accept" or "Decline". If the Family Medicine clinician clicks "Decline" then a reason must be given for declining. If the clinician decides a referral is appropriate, he/she clicks "Accept" and informs the patient that she will be contacted by CTIS. The referral is also included in the patient instructions. Within one week, a CTIS counselor will receive the referral through EPIC/EMR, and contact the patient.

When the patient is contacted by the CTIS Pregnancy Health Information specialist, a brief patient interview will be conducted with a risk assessment and counseling regarding the medication and potential effects if the patient were to become pregnant, using the standard of care practices that are currently used for all callers to the CTIS Pregnancy Health Information Line. The patient will also be given information about contraception, efficacy of rates of each contraceptive method and the safety of each method based on the USMEC guidance for the patient's medical condition. She will be instructed that she can return to her Family Medicine clinician for contraceptive service delivery. She will also be offered a referral to Reproductive Medicine at UCSD for further counseling if desired/necessary. The referring Family Medicine clinician will be informed of the outcome of the referral via an EMR report. This report will include the USMEC contraceptive guidance for the patient's medical condition.

After the counseling is completed, the patient will be asked if she is interested in participating in the research study. If the patient does not consent to participate in the study, she will still receive the counseling and an EMR report will still be sent to her referring provider but she will not be contacted at a later time regarding her contraceptive utilization.

If the woman decides that she is interested in participating in the research study, she will be orally consented by CTIS Pregnancy Health Information Line Research Assistant in the Department of Pediatrics at UCSD. If the patient consents to participation, she will be contacted one week, one month and three months after the initial telephone interaction and asked several questions regarding her current contraceptive utilization and any changes from the time of the last interview. Upon completion of the three-month follow-up, participants will also be asked to complete a satisfaction survey.

ELIGIBILITY:
Inclusion Criteria:

1. Age of participants: 18-45 years old
2. Gender of participants: Female
3. Ethnic Background: No limitation, will include minorities and Spanish speaking participants
4. Health Status: no limitation
5. Sexually active with men

Exclusion Criteria:

1. Currently Pregnant
2. Not sexually active with men
3. History of hysterectomy
4. Removal of both ovaries

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2012-01-05 (Actual); Primary Completion 2013-10-30 (Actual); Study Completion 2015-09-22 (Actual)

PRIMARY OUTCOMES:
Change in Contraception Utilization | one week, one month, three months
  Does specialized counseling improve (change) the utilization of more effective contraception among women in this population. We will measure the change in contraception utilization via a survey that participant will complete at each time frame.

SECONDARY OUTCOMES:
Proportion of women identified through Electronic Medical Record who are able to be contacted of Electronic Medical Record Referral | one week
  Can an electronic medical record referral to a Teratogen Information Line facilitate access to specialized counseling on the medication and effective contraception. We will measure the feasibility of the Electronic Medical Record Referral by assessing how many referrals are requested and how many referrals successfully result in teratogen/contraception counseling.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Mody, MD MPH, Study Director — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

REFERENCES:
- [Derived] Mody SK, Wu J, Ornelas M, Kernahan C, Salas E, Kao K, Felix R, Chambers C. Using the electronic medical record to refer women taking category D or X medications for teratogen and contraceptive counseling. Birth Defects Res A Clin Mol Teratol. 2015 Jul;103(7):644-7. doi: 10.1002/bdra.23396. Epub 2015 Jun 23. PMID 26100297